CLINICAL TRIAL: NCT03450382
Title: Hans Kai: Impact of a Peer Lead Community Health Program on Behavior Change, Mental Health, Health Efficacy and Social Support Comparative Control Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: New Principal Investigator
Sponsor: NorWest Co-op Community Health (Other)
Responsible Party: Principal Investigator, Mike Sadlowski, Health Promoter, NorWest Co-op Community Health
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 02222018
Record Dates: First submitted 2018-02-22; First posted 2018-03-01 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2018-02

CONDITIONS: Health Behavior
Keywords: community health; mental health; behavior change; social support; health promotion
MeSH Terms: conditions — Health Behavior; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Open label, quasi-experimental clinical trial comparative study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hans Kai Participant (Experimental): Participants receiving Hans Kai intervention
  Interventions: Other: Hans Kai Education
- Control (No Intervention): Participants not enrolled in Hans Kai

INTERVENTIONS:
Other: Hans Kai Education — 9 weeks of health education classes preceding social group formation into Hans Kai. Peer led support focused on behavioural change.
  Arms: Hans Kai Participant

SUMMARY:
To study the difference between participants interested in a lifestyle change when enrolled in Hans Kai or not when comparing behaviour change, social support, self health efficacy and mental health. Hans Kai is a community based, peer led program that is low cost and self sustaining, which places participants through a 9 week health school to learn skills related to improving health such as nutrition, exercise, sleep, stress management etc. Once completed, participants form a Hans Kai group and continue meeting independently of health care providers

DETAILED DESCRIPTION:
Research Question Does Hans Kai have a greater influence on healthy behavior change, mental health status, social connectedness, and self-health efficacy outcomes compared to community healthcare clients with access to health education programming.

Hypothesis - Hans Kai members will experience higher mental health improvement scores compared to control group.

Hans Kai members will experience greater social connectedness compared to control group.

Hans Kai members will experience greater self-health efficacy compared to control group.

Hans Kai members will adopt more behavior changes compared to control group.

Null Hypothesis - There is no significant difference between Hans Kai members and control group in terms of mental health improvement scores.

There is no significant difference between Hans Kai members and control group in terms of social connectedness scores.

There is no significant difference between Hans Kai members and control group in terms of self-health efficacy scores.

There is no significant difference between Hans Kai members and control group in terms of adopted behavior change numbers.

In order to meet the demand for health programming in and reduce the prevalence of chronic disease NorWest developed the HANS KAI Project. Hans Kai is a self-sustaining, participant led health program for individuals wanting to maintain or improve their health. Hans Kai groups consist of 8-40 people per group in communities or workplaces. Hans Kai empowers individuals to take control of their own health and provides a unique opportunity for participants to have an active role in improving or maintaining their own health and well-being and that of their community.

HANS Kai Focuses on a number of factors relating to health including:

Healthy eating, physical activity, managing sleep and stress, mental health, physical health indicators, leadership and social supports. The program is participant led which enables members to have an active role in their health and the health of their families and communities.

Currently NorWest has trained 37 people in 5 provinces across Canada to deliver HANS KAI in their community and demand is growing. NorWest has developed a Teen and Family HANS KAI to address health across the ages.

HANS KAI's initial research phase assessed roughly 60 participants over 2 years to determine the impact of Hans Kai on strategic health indictors and influences. Our research and evaluation showed statistically significant improvements in:

Mental Health (prior to HANS Kai 33% had Flourishing Mental Health at 12 months 69% had Flourishing Mental Health) Physical Activity Knowledge of Health Connection to Resources Increased Social Connections, and Upward trends in nutrition. As the program continued to evolve, community members and participants were involved in every phase, giving community feedback on important health related topics they wanted discussed and to be given more information on. This lead the researchers toward the second phase of research which now focuses heavily on behavior change. Putting into practice the information that participants learn was the highest feedback received, and this echoes trends in health promotion interventions, as preventative healthcare and integrated service becomes the pinnacle to healthy communities. Empowering people and building their resilience is dependent on needs and perceived value of different lifestyle influences. For instance, an economically disadvantaged family may struggle on a low income, but may find value in the Hans Kai nutrition classes on how to feed their family healthy options and recipes on a fixed budget. Addressing a change from eating take-out to home cooking helps to move this family towards better health and become economically stronger through education and application. Building on this scenario, Hans Kai also serves to bolster social engagement, drawing out isolated individuals to engage in their communities, increasing their mental health and well-being. The researchers strive to prove that this support carries over into the overall lifestyle, increasing the likelihood and motivation to improve physical activity levels with other group members interested in the same. This increase in self-efficacy promotes community and family leadership, as others see positive life choices, they are likely to join in, seeing family walks become routine and volunteering in community engagement on the rise.

The researchers are wanting to prove that community led health programs lead to health behaviour changes in healthy lifestyle choices with social support and self-efficacy.

After completing our first phase of research, the researchers were able to determine challenges and how to improve them as research heads into the second phase. Creating group champions to help collect interval research data and modifying our research to determine a power difference between a control and Hans Kai member was of the utmost importance. The research objectives will be looking to discover the differences between non Hans Kai community members and Hans Kai members in the areas of: self-efficacy, behavior change, physical activity, nutrition, mental health and community connectedness. Data comparisons from initial baselines without the Hans Kai intervention, followed by a 9 week survey after Hans Kai participants have completed the health school, followed by a 6 month and one year survey will be assessed. The purpose in completing these objectives is to determine whether the Hans Kai model produces better results in each of the mentioned areas for participants interested in a lifestyle change compared to those participants not introduced to the Hans Kai concept of education. If successful, the Hans Kai model will be further studied and promoted to more community health clinics as a low cost method to produce positive healthy behaviours to communities.

ELIGIBILITY:
Inclusion Criteria: Participants must be committed to making a lifestyle change

-

Exclusion Criteria:

* cognitively impaired
* Under 18
* students of children of Research team
* clients in emergency/life threatening conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Behaviour Change | 1 year
  To determine the power difference between Hans Kai participants and control group with respect to behavior change. Readiness to Change, Confidence to Change Questionnaire: Gillespie & Lenz (2011) will be used to measure this outcome.
Self-health Efficacy | 1 year
  To determine the power difference between Hans Kai participants and control group with respect to self-health efficacy. Health Self-Efficacy Questionnaire: Lee, Hwang, Hawkins & Pingree (2008) will be used to measure this outcome.
Social Support | 1 year
  To determine the power difference between Hans Kai participants and control group with respect to Social Support. A Social Connectedness Questionnaire developed by researchers will be used to measure this outcome.
Mental Health | 1 year
  To determine the power difference between Hans Kai participants and control group with respect to mental health. Mental Health Questionnaire: Keyes, C.L.M. (2009) will be used to measure this outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Leanne LeClair, PHD, Study Director — University of Manitoba
Locations (1):
- Access NorWest, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.